CLINICAL TRIAL: NCT06150872
Title: Early Feasibility Study to Evaluate the Safety of Photochemical Tissue Passivation (PTP) Treatment of Saphenous Vein Grafts in Participants Undergoing Elective CABG
Brief Title: Photochemical Tissue Passivation Treatment of Saphenous Vein Grafts in CABG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DurVena, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUR-001
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
Keywords: saphenous vein grafts; CABG surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Each subject will have at least 2 saphenous vein grafts. One graft will be randomized to treatment and one graft will be randomized to control. The outcomes assessor will be blinded to which graft has been treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Photochemical tissue passivation group (Experimental): Photochemical tissue passivation of a saphenous vein graft
  Interventions: Device: DurVena Photochemical Tissue Passivation
- Standard of care group (No Intervention): Standard of care treatment of a saphenous vein graft

INTERVENTIONS:
Device: DurVena Photochemical Tissue Passivation — Treatment of a saphenous vein graft with the DurVena Photochemical Tissue Passivation device.
  Arms: Photochemical tissue passivation group

SUMMARY:
Early feasibility study of the DurVena Photochemical Tissue Passivation (PTP) device for treatment of saphenous vein grafts in participants undergoing elective coronary artery bypass graft (CABG) surgery. Study to be conducted outside the U.S.

DETAILED DESCRIPTION:
The Photochemical Tissue Passivation (PTP) treatment of a saphenous vein graft (SVG) is indicated for the reduction of intimal hyperplasia and graft failure rate in SVGs after coronary bypass graft (CABG) surgery. The primary study objective, in this early feasibility study outside the US, is to characterize the safety profile of the PTP device when used during CABG surgery in participants with multivessel atherosclerotic coronary artery disease (CAD).

This is a prospective, randomized, within-subject controlled early feasibility study.

Up to 15 participants with multivessel CAD will be recruited for this study and followed for a minimum of 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation.
2. Age 21 years or older.
3. Planned and scheduled on-pump, arrested heart CABG.
4. Two or more vein grafts to native vessels having at least 75% stenosis and comparable runoff.
5. IMA graft indicated for the LAD.
6. Appropriately sized and accessible target coronary arteries, with a minimum diameter of 2 mm and adequate vascular bed (without significant distal stenosis), as assessed by pre-operative cardiac angiography and verified by diameter gauging intraoperatively.

   -

Exclusion Criteria:

1. Concomitant non-CABG cardiac surgical procedure.
2. Prior cardiac surgery.
3. Emergency CABG surgery (e.g., cardiogenic shock, inotropic pressure support, intraaortic balloon pump, ECMO).
4. Contraindication for on-pump CABG with cardioplegic arrest (e.g., severely calcified aorta).
5. Calcification at the intended anastomotic sites, as assessed upon opening of the chest and before randomization.
6. Platelets < 50,000/mm3 or other evidence of coagulopathy, INR greater than 1.5 in the absence of anticoagulation therapy.
7. Infection (WBC ≥12.5 x 103/ml and or temperature ≥100.5°F/38°C).
8. History of cerebral vascular accident (CVA) or transient ischemic attacks (TIA) within the last 3 months.
9. Unwilling or unable to receive blood transfusion.
10. Inability to undergo treatment with heparin.
11. Participants on dialysis or GFR of <30 ml/min/1.73m2.
12. Primary liver disease with bilirubin, SGOT, or SGPT > 4X upper limit of normal.
13. Prior history of allergic reaction to contrast media with anaphylaxis or severe peripheral edema.
14. Any medical condition that, in the opinion of the investigator, would compromise the safety of the participant or quality of the study data.
15. Pregnancy and nursing or lactating.
16. Current, or past participation in a clinical trial within the past 30 days.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Major cardiac adverse events (MACCE) | 30-days
  Major adverse cardiac and cerebral events (MACCE) including all-cause mortality, MI, stroke, and revascularization

SECONDARY OUTCOMES:
Major cardiac adverse events (MACCE) | 6-months
  Major adverse cardiac and cerebral events (MACCE) including all-cause mortality, MI, stroke, and revascularization
Major cardiac adverse events (MACCE) | 1-year
  Major adverse cardiac and cerebral events (MACCE) including all-cause mortality, MI, stroke, and revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Abdusalom Abdurakhmanov, MD, Principal Investigator — Republican Scientific Center of Emergency Medical Care, Uzbekistan
Locations (1):
- Republican Scientific Center of Emergency Medical Care, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No